CLINICAL TRIAL: NCT01261065
Title: Mechanisms of Improvement With Beta-Blocker Treatment in Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Biykem Bozkurt, MD, Michael E. DeBakey VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VA-CDA
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Cardiomyopathy
Keywords: beta blockers; heart failure; contractility; remodeling
MeSH Terms: conditions — Heart Failure; Cardiomyopathies | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: carvedilol — Patients with heart failure and LVEF < 35 % were treated with maximally tolerated dose of carvedilol for a period of six months. Target dose was 25 mg bid or 37.5 mg bid if patient's baseline weight > 80 kg.
  Other Names: coreg

SUMMARY:
The overall hypothesis of this application is that the improvement in LV ejection performance following treatment with betablockers is due, at least in part, to improvement in intrinsic myocardial contractility.

DETAILED DESCRIPTION:
The immediate specific objectives of this application are two-fold: (1) to determine whether the observed improvement in LV ejection performance is due to alterations in intrinsic cardiac myocardial contractility and (2) to determine whether changes in LV contractile reserve following an infusion of intravenous milrinone can be used to predict a salutary response to beta-blockers. The immediate specific objectives of this proposal will be addressed in the following two Specific Aims: In Specific Aim 1, we will determine whether the observed improvement in LV ejection fraction following treatment with beta-blockers is due to changes in intrinsic myocardial contractility, as opposed to changes in LV remodeling (i.e. reduction in LV volume) or changes in LV loading conditions. Changes in LV function will be evaluated using proven indexes, one an ejection phase index: the relation of end-systolic stress (ESS) to the mean velocity of fiber shortening (VCF), considered a relatively load independent measure of contractility. Changes in LV structure will be evaluated using echocardiography. In Specific Aim 2, we will determine whether the salutary response to beta-blockers can be predicted by measuring "contractile reserve", defined as a change in contractility determined by the relation of the mean velocity of fiber shortening (VCF) to end-systolic stress (ESS) in response to intravenous milrinone infusion at the cardiac catheterization lab prior to the institution of beta-blockade. The response to treatment with beta-blockers will be assessed by measurement of LV ejection fraction and LV end-diastolic volume by echocardiography after 6 months of treatment with beta-blockers, and these measurements will be correlated with the respective changes in contractile reserve measurement at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older.
2. Man or nonpregnant women (only women who are postmenopausal, surgically sterile or practicing an acceptable method of contraception)
3. Patients with dilated nonischemic cardiomyopathy with LVEF< 35% and NYHA Class III-IVa heart failure
4. Patients on standard stable medical therapy with Ace inhibitors (or hydralazine and nitrates or Angiotensin II Receptor blockers if Ace-intolerant), diuretics and or digoxin for at least 1 month prior to enrollment in the study.
5. Heart failure symptoms have to be present for at least 3 months
6. Written informed consent

Exclusion Criteria:

1. Ischemic heart disease documented by cardiac catheterization with any coronary obstructive lesion > 50% stenosis, history of myocardial infarction, coronary artery bypass surgery , percutaneous coronary angioplasty or stenting
2. Uncorrected primary valvular disease, obstructive or restrictive cardiomyopathy.
3. Systolic blood pressure >170 or <85 mm Hg or diastolic blood pressure >100 mm Hg; heart rate <50 bpm.
4. Sick sinus syndrome or advanced heart block (unless treated by a pacemaker), symptomatic or sustained ventricular tachycardia not controlled by antiarrhythmic drugs or an implantable defibrillator
5. Cor pulmonale, obstructive pulmonary disease requiring oral bronchodilator or steroid therapy
6. Active malignancy, or a systemic or terminal disease that would limit physical function or survival during the trial
7. Active and known drug or alcohol dependence or any factors that will interfere with the study conduct or interpretation of results.
8. Clinically important hepatic or renal disease; or any condition other than heart failure that could limit survival
9. Platelet count <100 000 mm3 or white blood cell count <3000 mm3, INR (international normalized ratio) >1.7
10. Current treatment with beta-blocker, beta-agonist, verapamil, chronic cyclic or continuous inotropic therapy, or use of an investigational drug within 30 days of entry into the challenge phase
11. History of drug sensitivity or adverse reactions to beta-blockers
12. Unwillingness to cooperate or give written informed consent, pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2001-12 (Actual); Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Load independent measure of contractility: Left ventricular velocity of circumferential shortening to left ventricular end systolic stress ratio | 6 months
  Mean velocity of circumferential fiber shortening (VCF) will be derived as = Left Ventricular Fractional shortening / Ejection Time.Left ventricular (LV) end-systolic stress will be calculated as = ([1.35 × P × LV endsysolic diameter]/(4 × LV posterior wall thickness in systole × (1+LV posterior wall thickness in systole /LV endsysolic diameter)))

SECONDARY OUTCOMES:
Left ventricular end diastolic and end systolic volumes, left ventricular end systolic stress, effective arterial elastance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Biykem Bozkurt, MD, Principal Investigator — Michael E.DeBakey VA Medical Center, Baylor College of Medicine
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bozkurt B, Bolos M, Deswal A, Ather S, Chan W, Mann DL, Carabello B. New insights into mechanisms of action of carvedilol treatment in chronic heart failure patients--a matter of time for contractility. J Card Fail. 2012 Mar;18(3):183-93. doi: 10.1016/j.cardfail.2011.11.004. Epub 2011 Dec 22. PMID 22385938